CLINICAL TRIAL: NCT06226181
Title: Amniotic Membrane for External Dacryocystorhinostomy and Comparison of Success Rate With Conventional Surgery for Patients With Nasolacrimal Duct Obstruction
Brief Title: Amniotic Membrane for Dacryocystorhinostomy
Acronym: AMDCRex
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CI-028-2017
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Nasolacrimal Duct Obstruction; Dacryocystorhinostomy
Keywords: Nasolacrimal Duct Obstruction; Dacryocystorhinostomy; Amniotic Membrane
MeSH Terms: conditions — Lacrimal Duct Obstruction | interventions — Dacryocystorhinostomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional dacryocystorhinostomy (Active Comparator): Patients undergoing conventional dacryocystorhinostomy using external approach.
  Interventions: Procedure: Conventional dacryocystorhinostomy
- Dacryocystorhinostomy using amniotic membrane (Experimental): Patients undergoing conventional dacryocystorhinostomy using external approach and adding amniotic membrane over the osteotomy, fixed with sutures.
  Interventions: Procedure: Dacryocystorhinostomy and amniotic membrane

INTERVENTIONS:
Procedure: Dacryocystorhinostomy and amniotic membrane — Dacryocystorhinostomy surgery with amniotic membrane placement on the osteotomy site.
  Arms: Dacryocystorhinostomy using amniotic membrane
Procedure: Conventional dacryocystorhinostomy — Conventional dacryocystorhinostomy surgery without adding amniotic membrane
  Arms: Conventional dacryocystorhinostomy

SUMMARY:
This study aims to compare the success rate of external dacryocystorhinostomy with and without amniotic membranes in patients with nasolacrimal duct obstruction.

DETAILED DESCRIPTION:
Naso-lacrimal duct obstruction (NLDO) causes epiphora, recurrent dacryocystitis, and skin fistulas. Its incidence increases with age. Dacryocystorhinostomy (DCR) is considered the standard treatment for NLDO. Authors describe similar success rates between external or endoscopic approaches. The former uses a skin approach, through which an osteotomy is made, allowing access to the lacrimal sac and subsequently to the middle meatus of the nasal cavity. On the other hand, endoscopic surgery uses an endonasal route to create a fistula towards the lacrimal sac, with the benefit of not generating visible scars in patients. The success of both surgeries depends on creating a wide osteotomy and the preservation of the mucosa around it, reducing the risk of scarring and stenosis of the ostium formed.

Some authors suggest that limiting the inflammatory process localized to the osteotomy may improve the surgical success rate. The use of mitomycin C (MMC) has been reported, with limited results due to variability in the concentration and methods of drug used.

Amniotic membrane (AM) has been used in ophthalmology, such as in pterygium surgery, chemical trauma, and inflammatory diseases of the ocular surface. In these contexts, AM limits the inflammatory response, promotes re-epithelialization, and reduces fibrosis. AM epithelial cells do not express HLA-A, B, C, or DR antigens on their surface, and therefore do not present a risk of rejection by the immune system.

This study aims to compare the success rate of external DCR with and without amniotic membranes in patients with NLDO.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Diagnosis of Nasolacrimal Duct Obstruction or Score ≥ 2 on the Munk Scale
* Patients able to undergo general anesthesia
* Patients able to keep follow-up
* Patients willing to participate in the study and signed informed consent

Exclusion Criteria:

* Patients with ocular surface diseases that affect surgical outcomes, such as blepharitis, lacrimal punctum epithelization, kissing punctae, facial nerve palsy, allergic conjunctivitis, etc
* Patients with eyelid malpositions
* Patients diagnosed with systemic inflammatory diseases, such as granulomatosis with polyangiitis, sarcoidosis, etc
* Previous history of facial trauma with nasal bone fractures
* Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Functional success rate | Pretreatment
  Clinical evidence of epiphora
Functional success rate | 1 day after surgery
  Clinical evidence of epiphora
Functional success rate | 1 week after surgery
  Clinical evidence of epiphora
Functional success rate | 3 weeks after surgery
  Clinical evidence of epiphora
Functional success rate | 3 months after surgery
  Clinical evidence of epiphora
Functional success rate | 6 months after surgery
  Clinical evidence of epiphora

SECONDARY OUTCOMES:
Osteotomy aspect | 1 day after surgery
  Endonasal aspect of osteotomy
Osteotomy aspect | 6 months after surgery
  Endonasal aspect of osteotomy
Nasolacrimal duct permeability | 1 week after surgery
  Permeability of nasolacrimal duct tested by canaliculi irrigation
Nasolacrimal duct permeability | 3 weeks after surgery
  Permeability of nasolacrimal duct tested by canaliculi irrigation
Nasolacrimal duct permeability | 3 months after surgery
  Permeability of nasolacrimal duct tested by canaliculi irrigation
Nasolacrimal duct permeability | 6 months after surgery
  Permeability of nasolacrimal duct tested by canaliculi irrigation
Visual acuity | Pre treatment
  Best corrected visual acuity
Surgical Complications | At the date of surgery
  Adverse events or unadvertised complications at the time of the surgery

OTHER OUTCOMES:
Visual acuity | 6 months after surgery
  Best corrected visual acuity

CONTACTS AND LOCATIONS:
Locations (1):
- Institiuto de Oftalmología Fundación Conde de Valenciana, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Woog JJ. The incidence of symptomatic acquired lacrimal outflow obstruction among residents of Olmsted County, Minnesota, 1976-2000 (an American Ophthalmological Society thesis). Trans Am Ophthalmol Soc. 2007;105:649-66. PMID 18427633
- [Background] Tooley AA, Klingler KN, Bartley GB, Garrity JA, Woog JJ, Hodge D, Bradley EA. Dacryocystorhinostomy for Acquired Nasolacrimal Duct Stenosis in the Elderly (>/=80 Years of Age). Ophthalmology. 2017 Feb;124(2):263-267. doi: 10.1016/j.ophtha.2016.10.018. Epub 2016 Dec 13. PMID 27986382
- [Background] Miranda Anta S, Blanco Mateos G, Valverde Collar C. [Dacryocystorhinostomy in adolescents and young adults]. Arch Soc Esp Oftalmol. 2011 Aug;86(8):243-6. doi: 10.1016/j.oftal.2010.12.014. Epub 2011 Jun 15. Spanish. PMID 21821190
- [Background] Huang J, Malek J, Chin D, Snidvongs K, Wilcsek G, Tumuluri K, Sacks R, Harvey RJ. Systematic review and meta-analysis on outcomes for endoscopic versus external dacryocystorhinostomy. Orbit. 2014 Apr;33(2):81-90. doi: 10.3109/01676830.2013.842253. Epub 2013 Dec 19. PMID 24354575
- [Background] Barmettler A, Ehrlich JR, Lelli G Jr. Current preferences and reported success rates in dacryocystorhinostomy amongst ASOPRS members. Orbit. 2013 Feb;32(1):20-6. doi: 10.3109/01676830.2012.747211. PMID 23387450
- [Background] Ali MJ, Psaltis AJ, Wormald PJ. Dacryocystorhinostomy ostium: parameters to evaluate and DCR ostium scoring. Clin Ophthalmol. 2014 Dec 9;8:2491-9. doi: 10.2147/OPTH.S73998. eCollection 2014. PMID 25525327
- [Background] Gonzalvo Ibanez FJ, Fuertes Fernandez I, Fernandez Tirado FJ, Hernandez Delgado G, Rabinal Arbues F, Honrubia Lopez FM. [External dacryocystorhinostomy with mitomycin C. Clinical and anatomical evaluation with helical computed tomography]. Arch Soc Esp Oftalmol. 2000 Sep;75(9):611-7. Spanish. PMID 11151233
- [Background] Liao SL, Kao SC, Tseng JH, Chen MS, Hou PK. Results of intraoperative mitomycin C application in dacryocystorhinostomy. Br J Ophthalmol. 2000 Aug;84(8):903-6. doi: 10.1136/bjo.84.8.903. PMID 10906101
- [Background] Nair AG, Ali MJ. Mitomycin-C in dacryocystorhinostomy: From experimentation to implementation and the road ahead: A review. Indian J Ophthalmol. 2015 Apr;63(4):335-9. doi: 10.4103/0301-4738.158082. PMID 26044474
- [Background] Arya SK, Bhala S, Malik A, Sood S. Role of amniotic membrane transplantation in ocular surface disorders. Nepal J Ophthalmol. 2010 Jul-Dec;2(2):145-53. doi: 10.3126/nepjoph.v2i2.3722. PMID 21505532
- [Background] Chavez-Garcia C, Jimenez-Corona A, Graue-Hernandez EO, Zaga-Clavellina V, Garcia-Mejia M, Jimenez-Martinez MC, Garfias Y. Ophthalmic indications of amniotic membrane transplantation in Mexico: an eight years Amniotic Membrane Bank experience. Cell Tissue Bank. 2016 Jun;17(2):261-8. doi: 10.1007/s10561-015-9540-7. Epub 2015 Dec 16. PMID 26675894
- [Background] Liu J, Sheha H, Fu Y, Liang L, Tseng SC. Update on amniotic membrane transplantation. Expert Rev Ophthalmol. 2010 Oct;5(5):645-661. doi: 10.1586/eop.10.63. PMID 21436959
- [Background] Nava-Castaneda A, Tovila-Canales JL, Monroy-Serrano MH, Tapia-Guerra V, Tovilla-Y-Pomar JL, Ordonez-Blanco A, Garnica-Hayashi L, Garfias-Becerra Y. [Comparative study of amniotic membrane transplantation, with and without simultaneous application of mitomycin C in conjunctival fornix reconstruction]. Arch Soc Esp Oftalmol. 2005 Jun;80(6):345-52. doi: 10.4321/s0365-66912005000600008. Spanish. PMID 15986275